CLINICAL TRIAL: NCT07242794
Title: The Effect of Podcast Use on Waste Management on Nursing Students' Knowledge Level and Satisfaction: A Randomized Controlled Trial
Brief Title: The Effect of Podcast Use on Waste Management on Nursing Students'
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Associate professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Podcast
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Waste Management; Satisfaction
Keywords: Nursing students
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: Control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Theoretical lectures and podcast listening
  Interventions: Other: Podcast listening
- Control (No Intervention): Theoretical lectures

INTERVENTIONS:
Other: Podcast listening — A podcast will be prepared to teach waste management to nursing students. Students will be able to listen to the podcast.
  Arms: Intervention

SUMMARY:
This study will be conducted to measure the effect of podcast use on waste management on nursing students' knowledge and satisfaction. The study was planned as a randomized controlled pretest-posttest study. The study sample will consist of 100 first-year students (50: Control; 50: Intervention) enrolled in the 2025-2026 Spring semester at Necmettin Erbakan University Faculty of Nursing. The study is planned to be conducted in February-March 2026 during the Spring semester of the 2025-2026 academic year. Data will be collected from first-year nursing students in a face-to-face classroom setting. Data will be collected using a "Personal Information Form," a "Waste Management Knowledge Test," and a "Satisfaction with Teaching Methods Survey." The data obtained from the study will be analyzed in a computer environment using SPSS (Statistical Package for the Social Sciences) version 22.0 (IBM Corp., Armonk, NY, USA). Data will be evaluated using descriptive statistics. The Kolmogorov-Smirnov test will be used to assess data for normal distribution. If data are normally distributed, the Independent Samples t-test will be used to compare two independent groups, the Paired Samples t-test will be used to compare two dependent groups, and the Pearson correlation will be used to compare the relationships between scales. If data are not normally distributed, the Mann-Whitney U test will be used to compare two groups.

DETAILED DESCRIPTION:
As with all healthcare professionals, student nurses may experience negative outcomes during clinical practice, such as infection transmission and sharps injuries. Proper waste disposal is crucial for the safety of patients and healthcare professionals, as is the knowledge level of both nurses and student nurses regarding waste management. Hospital-acquired infections can be prevented through medical waste management. It is equally important for nurses to be knowledgeable about preventing hospital-acquired infections. Equally important, student nurses should receive training in this area. Descriptive studies on waste management among nursing students have identified a lack of knowledge about waste management, and demographic characteristics (such as age, gender, and waste management training) influence their knowledge levels. The literature review found no studies other than descriptive studies on waste management. Student nurses are more likely to encounter problems such as infection transmission or sharps injuries when they first enter clinical practice. Waste management is crucial for student nurses to avoid these problems. Unless waste management is properly learned and implemented, patients and all healthcare professionals may be exposed to infectious infections such as hospital-acquired infections. To protect human and environmental health, waste management should be taught and practiced from the first year of nursing onward. Podcasts allow for the reach of a very wide audience. Podcast use is increasing in undergraduate nursing education. However, there is still a lack of literature evaluating the impact of podcast use in health education. It has been found that using topic-appropriate podcasts in undergraduate nursing education increases the knowledge and practical skills of nursing students. Podcats are an effective, innovative, and cost-effective learning technique for social interaction. The use of podcasts as a learning technique in health education has resulted in behavioral changes and increased satisfaction. In a study using podcasts in conjunction with a different learning technique, nursing students were asked to listen to a podcast before class using a flipped classroom method. This study observed that the use of podcasts in learning supports flexibility in education.

ELIGIBILITY:
Inclusion Criteria:

* Taking the Fundamentals of Nursing course for the first time.
* Voluntarily participating in the research.

Exclusion Criteria:

* Having graduated from a Health Vocational High School or having previously taken the
* Fundamentals of Nursing course,
* Having difficulty understanding and speaking Turkish,
* Not attending the theoretical training on the day of the waste management course,
* Having hearing loss, requiring the use of hearing aids, or having a condition that prevents the use of headphones,
* Not having the necessary equipment (phone, headphones, or internet access) to listen to the podcast content,
* Not attending the podcast event.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Waste management information | Up to 1 month
  Nursing students' waste management knowledge levels will be determined. The "Waste Management Knowledge Test," developed by the researchers, will be used for this purpose.

SECONDARY OUTCOMES:
Satisfaction with the teaching method | Up to 1 month
  Nursing students' satisfaction with learning by listening to podcasts will be determined. A "Satisfaction with Teaching Methods Survey" developed by the researchers will be used for this purpose.

IPD SHARING:
Plan to Share IPD: No